CLINICAL TRIAL: NCT02165423
Title: Discharge to Home and Chronic Illness Care Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Stacee Lerret, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: CHW 14/66
Record Dates: First submitted 2014-06-12; First posted 2014-06-17 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Solid Organ Transplant
Keywords: pediatric; solid organ transplant; parents; heart; kidney; liver

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Experimental): Ten parents will be randomized to the control group defined as 'usual care' and ten to the intervention group, stratified by type of transplant.
  Interventions: Behavioral: myFAMI iPad application
- Intervention (Experimental): Ten parents will be randomized to the control group defined as 'usual care' and ten to the intervention group, stratified by type of transplant.
  Interventions: Behavioral: myFAMI iPad application

INTERVENTIONS:
Behavioral: myFAMI iPad application

SUMMARY:
The purpose of this study is to address a gap in knowledge needed for care of children with solid organ transplantation (SOT) and their parents by combining mHealth technology with an individualized family centered self-management intervention (referred to as myFAMI). This study is critical to the increased understanding of hospital to home transition and family management at home with the potential to transform the way clinicians approach the care of complex chronic illness children and families.

ELIGIBILITY:
Inclusion Criteria:

* parent's child has undergone a heart, kidney, or liver transplant and is being discharged home from the hospital
* the parent is English speaking (to date the tools being used have been validated for English participants only)
* parent is 18 years of age or older
* patient is 17 years of age and younger.

Exclusion Criteria:

* presence of significant communication or cognitive impairment on the part of the parent that would preclude completion of questionnaires based on self-report
* parent and child has experienced the discharge to home transition from a previous transplant.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of myFAMI on 30-day post-discharge outcomes. | 30 days following enrollment
  Hypothesis: Compared to parents who received standard discharge preparation (usual care), parents receiving myFAMI will report:
  i) Better care coordination, ii) Higher quality of discharge teaching, iii) Greater readiness for hospital discharge, iv) Improved post-discharge coping, v) Improved family functioning, vi) Better self-management of medication and treatment regimens vii) Fewer emergency department visits and hospital readmissions

SECONDARY OUTCOMES:
Examine the acceptability of myFAMI: | Enrollment plus 30 days
  2. Examine the acceptability of myFAMI: The content of the interview will focus on strengths and weaknesses of iPad® technology in preparing parents for hospital discharge utilizing both survey and qualitative questions

CONTACTS AND LOCATIONS:
Overall Officials: Stacee Lerret, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States